CLINICAL TRIAL: NCT01740752
Title: Enhancing Treatment for Adult Anorexia With a Couple-Based Approach
Brief Title: UCAN2: Uniting Couples in the Treatment of Anorexia Nervosa
Acronym: UCAN2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11-1990; 1R01MH093615-01A1 (NIH)
Record Dates: First submitted 2012-11-08; First posted 2012-12-04 (Estimated); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; eating disorder; couples; relationships; couple therapy
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- UCAN+CBT (Experimental): This condition includes 22 UCAN sessions and 22 CBT sessions, totaling 44 psychotherapy sessions. UCAN is a manualized, 22-session Cognitive Behavioral Couple Therapy (CBCT) intervention that engages the couple to target the core psychopathology of AN and address the uniquely challenging stress that AN places on intimate relationships. The CBT proposed for this study is a 22 session adaptation of the manualized intervention that has been employed successfully as an outpatient post-hospitalization therapy and in an National Institute of Mental Health multisite study of fluoxetine with elements from the CBT manual used in McIntosh et al (PubMed 15800147).
  Interventions: Behavioral: UCAN+CBT
- CBT (Experimental): In this condition, participants will receive a higher "dose" of individual CBT, with 44 total sessions. Our experience with patients in the pilot strongly suggests that a higher dose of CBT will allow for further, fruitful discussion and exploration of key individual issues and is unlikely to be experienced as diluted or a slow approach to treatment. Most of these patients have complicated histories, long-standing eating disorders, and complex comorbid conditions.
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: UCAN+CBT — weekly manualized couple therapy plus weekly manualized individual CBT
  Other Names: CBCT
  Arms: UCAN+CBT
Behavioral: CBT — weekly manualized higher "dose" of individual CBT
  Arms: CBT

SUMMARY:
Uniting Couples in the treatment of Anorexia Nervosa (UCAN2) is a collaborative treatment research study between the University of North Carolina (UNC) Eating Disorders Program and the UNC Department of Psychology and is funded by the National Institute of Mental Health. The study examines two comprehensive treatments as couples face the challenges of anorexia nervosa (AN). The program helps patients with AN and their partners address AN symptoms and unique stresses that AN places on the romantic relationship.

DETAILED DESCRIPTION:
No single, conventional treatment has been shown to significantly benefit adults with AN, which ranks among the leading causes of disability and premature death in young women. The investigators propose to test the hypothesis that a novel, couple-based intervention developed for adult AN (UCAN) significantly enhances treatment outcome and reduces risk of relapse compared with treatment conducted entirely on an individual basis, the standard mode of treatment delivery in the community. The investigators plan to compare UCAN with individual treatment in a randomized controlled trial (RCT). All participants with AN will receive a common set of core interventions, including medical management, nutrition counseling, and a base level of individual cognitive-behavioral therapy (CBT), with randomization either to: 1) UCAN couple-based intervention or 2) a higher "dose" of individual CBT. The partners are involved in varying ways and to varying degrees in treatment. In addition, progress will be followed for one year after completion of active treatment.

ELIGIBILITY:
Inclusion Criteria

1. Participant with AN must have:

   1. Current Diagnostic and Statistical Manual of Mental Disorders Fourth Edition (Text Revision) (DSM-IV-TR) criteria for AN, restricting or binge/purge subtype; BMI between 15.0-19.0 currently or sometime in the past 3 months.
   2. Adequate insurance coverage to support a higher level of care including but not limited to partial hospitalization or inpatient treatment.
2. Both members of couple must be:

   1. At least 18 years of age.
   2. English speaking.
   3. Involved in a committed relationship for at least 6 months, regardless of sexual orientation.
   4. Wiling to participate in treatment.

Exclusion Criteria

1. Participant with AN cannot be: Unwilling to suspend other treatment for AN for the duration of the study.
2. Partner cannot meet: Current DSM-IV-TR criteria for AN, restricting or binge/purge subtype. We will exclude couples in which both partners have a diagnosis of AN.
3. Neither member of couple can have:

   1. Alcohol or drug dependence in the past year.
   2. Current significant suicidal ideation (from interview or depression assessment).
   3. Severe depression that would seriously interfere with functional capacity, as judged by the PIs or study physician.
   4. Developmental disability that would impair the ability to benefit from the intervention.
   5. Any psychosis, schizophrenia, or bipolar I disorder, unless stably remitted on maintenance therapy for at least 1 year.
   6. Moderate to high levels of physical violence from participant/partner as reported during baseline interview.
   7. Previously participated in the UCAN couple treatment condition in the preliminary couples treatment study (#07-1429. UCAN: Uniting Couples (in the treatment of) Anorexia Nervosa)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-07 (Actual); Primary Completion 2019-01-17 (Actual); Study Completion 2019-01-17 (Actual)

PRIMARY OUTCOMES:
Change in Body Mass Index (BMI) from baseline through 12 month follow-up | BMI is measured at baseline, weekly during the first 6 months (while in active treatment), and at each time point through 12 month follow-up
  BMI is a measure of body fat based on height and weight that the study is using to track weight changes throughout the course of the study. In AN, weight loss indicates the severity of the disease and weight gain is associated with recovery. Therefore, BMI is used to track progress in recovery.
Change in Global Eating Disorder Examination (EDE) Scores from baseline through 12 month follow-up | The EDE is assessed at baseline and each time point from end-treatment through the 12 month follow-up
  The EDE measures the frequency in which a patient engages in behaviors indicative of an eating disorder over a 28 day period.

SECONDARY OUTCOMES:
Dropout (the percentage of individuals who withdrew participation from treatment) | Month 6/ end-treatment assessment
  Dropout will be compared in the two treatment groups to see if a certain intervention enhances compliance with treatment.
Treatment satisfaction scores as measured with the Client Satisfaction Questionnaire (CSQ) | Month 6/ end-treatment assessment
  Treatment satisfaction is measured at end-treatment with CSQ. The CSQ rates effectiveness of, and satisfaction with services received.
Relationship satisfaction as measured with the Dyadic Adjustment Scale (DAS) and DAS-4 | Baseline through 12 month follow-up. Also, all patients and partners in the UCAN + CBT group only rate relationship satisfaction weekly (up to 23 weeks) during active treatment.
  Extent to which someone is happy in his or her relationship.

OTHER OUTCOMES:
Cost effectiveness ratio (is the ratio of the change in costs to incremental benefits of a therapeutic intervention or treatment) | Cost effectiveness is measured at each time point from 3 month follow-up to 12 month follow-up
  The cost effectiveness ratio will be calculated using utilization data from the McKnight Follow-up of Eating Disorders (MFED).

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Bulik, PhD, Principal Investigator — UNC Chapel Hill Department of Psychiatry; Donald Baucom, PhD, Principal Investigator — UNC Chapel Hill Department of Psychology
Locations (1):
- UNC Center of Excellence for Eating Disorders, Chapel Hill, North Carolina, United States